CLINICAL TRIAL: NCT02158455
Title: No-touch Saphenous Vein Grafts vs Radial Artery Grafts; A Randomized Trial.
Brief Title: Vein vs Arterial Grafts for Coronary Artery Bypass Grafting Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Mats Dreifaldt, MD PhD, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTSVGRA
Record Dates: First submitted 2014-04-30; First posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Angina Pectoris
Keywords: CABG; Saphenous vein; Radial artery
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NT SVG grafts (Experimental): NT SVG randomized for revascularization of left or right coronary territory
  Interventions: Procedure: NT SVG grafts
- RA grafts (Active Comparator): RA grafts randomized for revascularization of left or right coronary territory
  Interventions: Procedure: NT SVG grafts

INTERVENTIONS:
Procedure: NT SVG grafts

SUMMARY:
The investigators have developed a novel technique for saphenous vein graft harvesting for coronary artery bypass grafting (CABG) where the graft is harvested with a pedicle of surrounding tissue. A randomized trial has shown a significantly higher patency rate for vein grafts harvested with this new methode compared to conventional harvesting technique 8.5 years after surgery (90 vs 76 %). In 2004 the investigators started a prospective randomized trial comparing patency between vein grafts harvested with surrounding tissue and radial artery grafts. The result showed that vein grafts harvested with surrounding tissue had a significantly higher patency rate compared to radial artery grafts 3 years after surgery (98 vs 84 %). The present study is a long-term follow-up (8 years) of the patients included in the second randomized trial. The hypothesis is that vein grafts harvested with surrounding tissue have a significantly higher patency rate compared to radial artery grafts 8 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Three vessel coronary artery disease

Exclusion Criteria:

* 65 years or older
* Elevated creatinine
* Raynauds disease
* Vein stripping

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Graft patency | 5 months
  The grafts will be categorized as either "open" or "closed". A stenosis of the graft exceeding 70 % of the lumen diameter will be considered as "closed".

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Örebro, Sweden